CLINICAL TRIAL: NCT05274698
Title: Efficacy Of Muscle Energy Technique On Shoulder Adhesive Capsulitis Post Mastectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samah Gameil Fakhry Serg, lecturer assistant of physical therapy ,Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003434
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Adhesive Capsulitis of Shoulder
MeSH Terms: conditions — Bursitis | interventions — Range of Motion, Articular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental group): (Experimental): This group includes 30 patients with adhesive capsulitis who will receive muscle energy techniques 1 session per day, 5 days a week for 8 weeks in addition to their conventional physical therapy program (Mobilization exercises, Posterior capsule stretching, and Range of motion exercises).
  Interventions: Behavioral: muscle energy technique; Behavioral: conventional physical therapy program (Mobilization exercises, Posterior capsule stretching, and Range of motion exercises) 1 session per day, 5 days a week for 8 weeks.
- Group B (Control group): (Other): This group includes 30 patients with adhesive capsulitis who will receive their conventional physical therapy program (Mobilization exercises, Posterior capsule stretching, and Range of motion exercises) 1 session per day, 5 days a week for 8 weeks.
  Interventions: Behavioral: conventional physical therapy program (Mobilization exercises, Posterior capsule stretching, and Range of motion exercises) 1 session per day, 5 days a week for 8 weeks.

INTERVENTIONS:
Behavioral: muscle energy technique — It is a manual treatment in which a patient produces a contraction in a precisely controlled position and direction against a counterforce applied by a manual therapist .Muscle energy techniques (MET) were originally developed to treat soft tissue, mobilize joints, stretch tight muscles and fascia, reduce pain and to improve circulation and lymphatic drainage.
  Arms: Group A (Experimental group):
Behavioral: conventional physical therapy program (Mobilization exercises, Posterior capsule stretching, and Range of motion exercises) 1 session per day, 5 days a week for 8 weeks. — Joint mobilization, specifically glenohumeral joint distraction, glenohumeral joint caudal glide, glenohumeral joint posterior glide, and glenohumeral joint anterior glide, will be applied with patients.
  Posterior capsule stretching will be applied with patients in side lying position. The scapula will be stabilized at the lateral side with the arm at 90° flexion. Stretching will be applied from the elbow with a downward force. The stretch will be repeated 10 times for 20 s each. A 30-s break will be given between each stretching .
  Range of motion exercises:
  Codman/ pendulum exercise ,Wall climbing exercise and Shoulder wheel exercise Circumduction of the shoulder joint clockwise and anticlockwise using shoulder wheel

SUMMARY:
The purpose of the study is to evaluate the effect of muscle energy technique on adhesive capsulitis post mastectomy.

DETAILED DESCRIPTION:
1. Subjects:

   Sixty patients who have adhesive capsulitis post- mastectomy will participate in this study .Their ages will range from 40 to 60 years. The participants will be selected from National Cancer Institute, Cairo University and randomly distributed into two equal groups.

   1.1 Design of the study:

   In this study the patients will be randomly assigned into two equal groups (30 patients for each group):

   1.1(a) Group A (Experimental group): This group includes 30 patients with adhesive capsulitis who will receive muscle energy techniques 1 session per day, 5 days a week for 8 weeks in addition to their conventional physical therapy program (Mobilization exercises, Posterior capsule stretching, and Range of motion exercises).

   1.1(b) Group B (Control group): This group includes 30 patients with adhesive capsulitis who will receive their conventional physical therapy program (Mobilization exercises, Posterior capsule stretching, and Range of motion exercises) 1 session per day, 5 days a week for 8 weeks.
2. Equipment:

2.1- Measurement equipment: 2.1.a-Visual analogue scale (VAS): The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain.

2.1.b-Goniometer :

One of the most common assessment methods is measuring range of motion (ROM) of the joint using a goniometer. This method has been used for almost 90 years. Baseline limitation on ROM of a patient can be obtained before treatment, and changes induced in this motion after therapeutic interventions is easily determined. Reliability studies on ROM measurement of the joint using goniometer have been studied in depth, and have shown high reliability 2.1.c-Shoulder Pain and Disability Index (SPADI):

Is a self-administered questionnaire that aims to measure pain and disability associated with shoulder disease .The Shoulder Pain and Disability Index (SPADI) was developed to measure current shoulder pain and disability in an outpatient setting. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability .

2. 2-Therapeutic equipment and tools: 3-Procedures of the study: 3.1-Measurement procedures: 3.1.a-A Visual Analogue Scale (VAS):

VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end, as illustrated in Fig. (1).The patient will mark on the line the point that they feel represents their perception of their current state. The VAS score will be determined by measuring in millimetres from the left hand end of the line to the point that the patient mark .

3.1.b- Goniometer: ( From supine lying position ,the measurements will be taken for shoulder flexion, abduction, and external rotation).

ELIGIBILITY:
Inclusion Criteria:

* • Female patients with age range between 40-60 years.

  * Shoulder ROM restriction.
  * Shoulder pain more than 3 months.
  * Patients with adhesive capsulitis abduction test and external rotation test positive.
  * Patients referral adhesive capsulitis with MRI

Exclusion Criteria:

* • Disease such as rheumatoid arthritis

  * Diabetes mellitus.
  * History of trauma or accidental injuries.
  * Neurological involvement (stroke, Parkinsonism, radiating pain to arm).
  * History of surgery on particular shoulder

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 2 month
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
Goniometer | 2 month
  ( From supine lying position ,the measurements will be taken for shoulder flexion, abduction, and external rotation).

OTHER OUTCOMES:
The Shoulder Pain and Disability Index (SPADI) | 2 month
  The SPADI consists of two dimensions (pain and disability) with a total of 13 questions. The pain dimension consists of five questions pertaining to the severity of an individual's pain. Disability will be assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living requiring the use of the upper extremities. To answer the questions, the patients will place a mark on a 10-cm VAS for each question. Verbal anchors for the pain dimension will be 'no pain at all' and 'worst pain imaginable' and those for the disability dimension were 'no difficulty' and 'so difficult it requires help'. Scores from both dimensions will be averaged to derive a total percentage score. Higher scores reflected more pain and greater disability

CONTACTS AND LOCATIONS:
Overall Officials: faculty of physical therapy, Study Director — teaching assistant of physical therapy cairo university
Locations (1):
- Faculty of Physical Therapy, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No